



### **TEEN ASSENT FORM (OPT: Program + Surveys)**

**IRB #:** 22811

**Study Title:** Project LIVE (Love, Inclusivity, Values, and Education)

Contact Information: Email: <a href="mailto:projectlive@unl.edu">projectlive@unl.edu</a> Phone: 515-410-6536

Website: https://go.unl.edu/projectlive

Social Media: @unl.projectlive on Facebook & Instagram

### **Key Information:**

- DMPS students registered at Hoover or All Points high schools and enrolled in Physical Education (P.E) classes at Hoover or a Learning Transition Period at All Points during the 2023-2024 school year are eligible to participate.
- Participation includes: 1 pre-test survey (30 minutes), 6 sessions of a sex trafficking prevention curriculum (45-minutes/session or 4.5 hours total), 6 post-session surveys (5 minutes each/30 minutes total), and 1 post-test survey (30 minutes). You are not being graded on the surveys.
- There are a few risks associated with this study (see below, page 2).
- Your information will be anonymous, and data may be shared (see below, page 2).
- You will have the chance to win a \$100 incentive for participating.
- You can get a copy of this form.
- Your participation is voluntary.

**Why are you being asked to be in this research study?** You are being asked to be in this study because you attend high school at either Hoover or All Points within the DMPS system during the 2023-2024 academic year and because you can understand spoken English.

**What will be done?** This study is aimed at preventing sexual exploitation of teens. The program will be given in your P.E. class. The two main parts of this project are:

- <u>Program Delivery:</u> The READY to Stand™ (RTS) Curriculum will be delivered in six 45-minute modules (e.g., healthy relationships, valuing self and others). The RTS curriculum will be presented to teens in English.
- <u>Program Evaluation</u>: You will be asked to take a survey before the curriculum is delivered (pre-test survey, 30 minutes), after each of the six sessions (post-session surveys, 5 minutes), and after all six sessions are complete (post-test survey, 30 minutes). These surveys are available in English and Spanish.

**What are the possible risks of being in this research study?** The risks to participation are minimal. When talking about topics like sex trafficking, people may sometimes feel sad,



anxious, or awkward. You can stop participating at any time or not answer any question(s) you don't want to answer. Also, you will be given a list of resources in Des Moines if you or someone you know needs help.

What are the possible benefits to you? Sometimes youth tell us that they enjoy participating in research and like to share their ideas and help other people and their community. However, you may not benefit from being in this project.

Will you be compensated for being in this research study? We will do a drawing for 1 in 5 \$100 gift cards for the surveys teens take before the program. We will do another drawing for 1 in 5 \$100 incentive for the surveys teens take after the program. Finally, we will also raffle a \$100 incentive at each of the 6 classes. There will be a total of 16, \$100 gift cards. We expect about 900 teens to participate so each teen has a 2% chance of winning a gift card. All teens will get project swag (e.g., bracelets, pencils). We will do the drawings within a few months of when you start this project. The person doing the drawing will be a researcher at UNL. They will do the drawing using a computer program to make sure it is fair and accurate. If you win a gift card, you will be asked to fill out a form saying you got the money. However, your survey answers/ feedback will not be connected to the form confirming receipt of the gift card.

How will information about you be protected? Reasonable steps will be taken to protect your privacy. What you tell us will be kept private. This means that we will not share what you tell us with other people UNLESS you tell us: (1) that you are being hurt or abused, (2) that you plan to hurt yourself or someone else, and/or (3) if someone else, like an elder or other teen or child, is being hurt or abused. If you tell us about these things and/or we were to witness these things, we will have to notify the Iowa Department Health and Human Services. We will also tell someone at your school like a counselor.

Finally, we will share your data, without any information that could identify you, like your name or where you live, in a special database for other scientists who are doing research. Sharing your data helps scientists learn new and important things more quickly. Any scientists interested in using your data would have to put in a special request, promise to keep your data safe, and promise not to try to learn your identity. We cannot remove your data if you change your mind because the data is anonymous. So, you are agreeing for your de-identified data (no names, etc.) to be put together with other teens' data to be shared in a database by saying you want to be in this study.

**Public Information About this Study.** ClinicalTrials.gov is a website that provides information about federally and privately supported clinical trials. A description of this clinical trial will be available (http://www.ClinicalTrials.gov) as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

What will happen if you decide not to be in this research study or decide to stop participating once you start? Participation is voluntary. You have the right to quit the study at any time or to not answer any question(s) that you do not want to answer. You will be entered to receive a gift card even if you refuse/skip questions on the pre-test/post-test/post-session survey or during the feedback session.



If you decide not to participate in this project, you will engage in an alternate health-related educational activity (if enrolled in P.E.) or an alternate activity typical for Learning Transition Period (such as independent reading, assignment/homework completion, etc.) supervised by your regular physical education teacher, Learning Transition Period teacher, or other school staff held in a different classroom than teens who are participating.

**Documentation of informed consent.** We will also inform your caregiver/legal guardian about this study and offer them the opportunity to withdraw you from any/all research activities. If you are over 18, your caregiver/guardian does not need to give you permission.

If you have any questions now or at any point during the study, please email (<a href="mailto:ProjectLIVE@unl.edu">ProjectLIVE@unl.edu</a>) or call (515-410-6536).

| Do you agree to participate? |
|------------------------------|
| YES |
| NO |
| Your Name: |
| Your School: |
| Your Grade in School: |
| Your Age: |
| Your Cell Phone Number: |
| Your Email: |
| Your Signature: |
| Date: |

The contact information is being collected solely for research purposes. We will never share this information.





## **GUARDIAN CONSENT FORM (OPT Programming and Surveys)**

Only legal guardians of youth younger than 18 and who attend HOOVER HIGH or ALL POINTS can complete this form.

- ✓ Guardians who return the form, whether it indicates their youth can or cannot participate, will receive a \$15 virtual VISA gift card.
- ✓ Youth who return the form, whether it indicates they can or cannot participate, will also receive a \$15 virtual VISA gift card.
- ✓ Deadline to sign and return:
  - o ALL POINTS: Friday, April 12, 2024
  - o HOOVER HIGH: Friday, April 12, 2024
- ✓ Please refer to PAGE 5 for signatures and return information!

**IRB** #: 22811

**Study Title:** Project LIVE (Love, Inclusivity, Values, and Education)

Contact Information: Email: projectlive@unl.edu Phone: 515-410-6536

Website: <a href="https://go.unl.edu/projectlive">https://go.unl.edu/projectlive</a>

Social Media: @unl.ProjectLIVE on Facebook and Instagram

### 1. Key Information:

- Des Moines Public Schools (DMPS) students registered at Hoover High School or All Points Academy during the spring, 2024 school semester are eligible to participate.
- Your teen's participation includes: 1 pre-test survey (30 minutes), 6 sessions of a sex trafficking prevention curriculum (45-minutes/session or 4.5 hours total), 6 post-session surveys (5 minutes each/30 minutes total), and 1 post-test surveys (30 minutes). Your teen will not be graded on the surveys.
- There are a few risks associated with this study (see below).
- Your teen's information will be anonymous (see below).
- Your teen's anonymous data may be shared (see below).
- Your teen will have the chance to win \$100 incentive for participating. This is in addition to the \$15 for returning this form.
- Your teen will be provided with a youth assent form and can decline to participate even if you say it is OK for them to participate.
- Please return by Friday, April 12, 2024.



**Invitation.** You are being asked to allow your teen to participate in a research project aimed at preventing sex trafficking of youth. The research is being conducted by Dr. Katie Edwards from the University of Nebraska-Lincoln, in collaboration with the Set Me Free Project and DMPS. The program will be incorporated into your teen's P.E. course (HOOVER students) or Learning Transition Period (ALL POINTS). The project is funded by the Centers for Disease Control and Prevention (CDC) and is not in response to any particular incident.

**Why is your teen being asked to be in this research study?** Your teen is being asked to be in this study because your teen attends either Hoover High School or All Points Academy during the winter/spring, 2024 academic semester.

What is the reason for doing this research study? DMPS wants to implement and receive feedback on READY to Stand™ (RTS) Curriculum, a school-based prevention program aimed at preventing sex trafficking. Beyond participating in the curriculum, we would like to get feedback from teens so that we can make the program as effective as possible for other youth.

**What will be done during this research study?** The project consists of the following elements.

- <u>Program Delivery</u>: The RTS Curriculum consists of six 45-minute modules (e.g., healthy relationships, valuing self and others), presented by trained Set Me Free Project Program Educators as a regularly scheduled part of your teen's PE or learning transition time classes. The RTS Curriculum will be presented to all teens in English.
- <u>Program Evaluation</u>: Your teen will be asked to complete a survey prior to program delivery (pre-test survey, 30 minutes), after each of the six sessions (post-session surveys, 5 minutes) and after all six sessions have been delivered (post-test survey, 30 minutes). There are no "wrong" answers on these surveys. Surveys will NOT be graded. They are anonymous. These surveys are available in English and Spanish.

How will my teen's data be stored or shared? We will protect the confidentiality of your teen's information to the extent possible. The surveys are anonymous and what your teen tells us will be kept private. This means that we will not share what they tell us with other people UNLESS they tell us: (1) that they are being hurt or abused, (2) that they plan to hurt themselves or someone else, and/or (3) if someone else, like an elder or other teen or child, is being hurt or abused. If you decide to allow your teen to participate in the project and your teen told us about any of these things or we were to witness child abuse, we will have to notify Iowa Department of Health and Human Services and someone in DMPS. We will also tell someone at your teen's school like a counselor.

Your teen's responses will be reported in terms of groups of participants rather than as individual cases. No names or other identifying information will be included.



Those who will have access to your teen's research records are the study personnel, the Institutional Review Board (IRB), and any other person, agency, or sponsor as required by law or contract or institutional responsibility. If these individuals were to access the data, your teen's name would not be associated with it.

Finally, the CDC has asked researchers to share as much data from this study as we can with other researchers. We will share your teen's data, without any information that could identify them in a special database for other scientists who are doing research. We will only share de-identified data, in which research participants and schools will be identified by a number, and DMPS will be referred to as "a school district in a city in the Midwest" (or a similar variation). Any scientists interested in using teens' data would have to put in a special request, promise to keep the data safe, and promise not to try to learn teens' identity. We cannot remove your teen's data if you change your mind because the data are anonymous. So, you are agreeing for your teen's de-identified data (no names, etc.) to be put together with other teens' data to be shared in a database by saying you want to be in this study. This sharing is not sharing your information for future research. It is only sharing data from this specific study.

**Public Information About this Study.** ClinicalTrials.gov is a website that provides information about federally and privately supported clinical trials. A description of this clinical trial will be available (http://www.ClinicalTrials.gov) as required by U.S. law. This website will not include information that can identify you or your teen. At most, the website will include a summary of the results. You can search this website at any time.

Certificate of Confidentiality. You should also know that we have a Certificate of Confidentiality from the Federal Government. This means that if someone came to us and asked for information about your teen or other people in the project, we could use this Certificate to refuse to give them information. This Certificate is to help us protect your teen's privacy. Yet, it does not prevent you or a member of your family from voluntarily releasing information about your teen or your teen's involvement in this research. If you give your written consent to someone to receive research information, then we may not use the Certificate to withhold information.

What are the possible risks of being in this research study? The risks to participation are minimal. Sometimes when talking about topics like sex trafficking, people may feel sad, anxious, or awkward. However, trained Program Educators and members of the research team will be available and accessible to teens during program implementation and data collection. We will also provide a list of resources they can access if they want help.

What are the possible benefits to your teen? Your teen may not benefit from being in this project. However, some people tell us that they enjoy participating in research and like to share their ideas and help other people and their community.

What are the possible benefits to other people? The benefits to society include a better understanding of how to prevent sex trafficking of teens.



What are the alternatives to being in this research study? Instead of being in this research study you can choose not to allow your teen to participate. If your teen does not participate, they will engage in an alternative activity (such as physical activity typical for teens enrolled in P.E. courses at Hoover High or regular classroom activities for those attending All Points Academy). Teens will be supervised by their regular teachers or other school staff if they do not participate in the RTS Curriculum.

What will being in this research study cost you or your teen? There is no cost to you or your teen to be in this research study.

Will your teen be compensated for being in this research study? We will do a drawing for 1 in 2 \$100 gift cards for the surveys teens take before the program; another drawing for 1 in 3 \$100 gift cards for the surveys teens take after the program. We will also raffle a \$100 incentive gift card after each of the 6 classes. For Spring, 2024 there will be a total of 8 \$100 gift cards. We expect about 175 teens to participate in spring, 2024 so each teen has a 4.5% chance of winning. All teens will get project swag (e.g., stickers, pencils). Drawings will be done electronically by a UNL researcher within a few months of the start of the program. If your teen wins a gift card, you will be asked to fill out a form saying the gift card was received, but your survey answers/feedback will not be connected to the form confirming receipt of the incentive. This is in addition to the \$15 virtual cards you and your teen will get for turning in this form.

What should you do if your teen has a problem during this research study? Your teen's well-being is important to us. If there is a concern as a direct result of being in this study, you should immediately contact Dr. Edwards listed at the beginning of this consent form. While participating in the study, your teen will receive and have ongoing access to a list of resources that they can contact. Also, participation is voluntary, and your teen can stop at any time or choose to not be involved, even if you say they can.

How will information about your teen be protected? All research records will be securely stored electronically through University-approved methods and will only be seen by the research team and/or those authorized to view, access, or use the records.

What are your teen's rights as a research subject? Your teen may ask any questions about this research and have those questions answered at any time. Your teen may also decide not to participate even if you say that they can participate. Your teen can stop participating at any time and can choose not to answer any questions and still be eligible for compensation.

Who should I contact if I have questions or concerns about this research project? If you have questions about this project, you can contact Dr. Katie Edwards, the principal investigator, by email (ProjectLIVE@unl.edu) or phone (515-410-6536). You can also contact the IRB at the UNL if you have questions at 402-472-6965 or irb@unl.edu.

What will happen if you decide not to allow your teen to be in this research study or decide they need to stop participating once they start? You can decide to allow your teen to be in this research study or not; you can have your teen stop being in this research study ("withdraw") at any time by emailing or calling us. Deciding not to allow your teen to be in



this research study or deciding to withdraw will not affect you or your teen's relationship with the investigator or with UNL. You and your teen will not lose any benefits to which you or they are entitled.

**Documentation of informed consent** You are voluntarily deciding whether or not to allow your teen to be in this research study. Please contact us if (1) you have read and **do not** understand this consent form and/or (2) you desire any element of the consent form clarified or explained to you. You can download this form at (Website: <a href="https://go.unl.edu/projectlive">https://go.unl.edu/projectlive</a>).

**Caregiver Consent Form.** I have read the information about the research being conducted by the University of Nebraska-Lincoln. Please check the box below indicating whether or not you want your teen to take part in programming and research.

| Place a check mark (X) in one of the boxes below. | | | | |
|---|---|---|---|---|
| | <b>YES</b> , my teen <b>has permission</b> to participate in the RTS program and associated research (pre-/post-surveys; post-session surveys). | | | |
| | <b>NO</b> , my teen <b>does not</b> have permission to participate in the RTS program or associated research (pre-/post-surveys; post-session surveys). | | | |
| Legal Guardian Information | | | | |
| Guardian/Parent Name (printed): | | | | |
| Guardian/Parent Signature: | | | Date: | |
| C 1' /D | | 1 | 1 44 F 1 . 1 | · C 12 |
| Guardian/Parent email: (a valid email must be provided to receive the \$15 virtual gift card) | | | | |
| Teen's Information | | | | |
| Teen's Name: | | | | |
| Teen's School:(check one) | | | Grade: | Teen's Age: |
| Ноо | ver All Points | | | |
| Toon's amail: (a | valid amail must be provided to receive | tha \$15 x | wirtual gift card) | |
| <b>Teen's email</b> : (a valid email must be provided to receive the \$15 virtual gift card) | | | | |

Please return this form by Friday, April 12, 2024

The form can be returned in any of the following ways, including:

- Returning to your teen's school (PE Teacher/Hoover, any teacher/All Points)
- Taking a picture of this signature page and emailing it to <a href="mailto:ProjectLIVE@unl.edu">ProjectLIVE@unl.edu</a>
- Taking a picture of the signature page and texting it to 515-410-6536
- Completing online: go.unl.edu/PLconsent23





#### SCHOOL PERSONNEL CONSENT F ORM

(District Wide Survey-all schools OTHER than Hoover and All Points)

IRB #: 22811

**Study Title:** Project LIVE (Love, Inclusivity, Values, and Education)

Contact Information: Email: <a href="mailto:projectlive@unl.edu">projectlive@unl.edu</a> Phone: 515-410-6536

Website: <a href="https://go.unl.edu/projectlive">https://go.unl.edu/projectlive</a>

Social Media: @unl.projectlive on Facebook & Instagram

# **Key Information:**

This is quick summary of the project:

- All school personnel working at any of the high schools in the Des Moines Public School (DMPS) system are invited to participate.
- Survey completion will take about 15 minutes.
- There are minimal risks associated with this study (as described below).
- Your de-identified data may be shared (as described below).
- You will be entered to receive a \$100 incentive for completing the survey.
- Your participation is voluntary.

**Invitation.** You are being asked to participate in a research project aimed at the prevention of sex trafficking of youth. The research is being conducted by Dr. Katie Edwards from the University of Nebraska-Lincoln, in collaboration with the Set Me Free Project and Des Moines Public School (DMPS) administrators and staff. The project is funded by the Centers for Disease Control and Prevention. It is important for you to know that this project is not in response to any particular incident.

**Why are you being asked to be in this research study?** You are asked to be in this study because you work in any high school/s in the DMPS system.

What is the reason for doing this research study? The purpose of this study is to prevent sex trafficking among teens in DMPS. School personnel (e.g., teachers, administrators, counselors, support staff) play an important role in this.

**What will be done during this research study?** To participate, you will complete a survey. You will answer questions about your perceptions of sex trafficking among



students, your role in prevention of sex trafficking among students, and some additional questions on attitudes and beliefs. There are no "wrong" answers to the survey; it will take about 30 minutes to complete.

**How will my data be stored or shared?** The surveys are confidential. Your responses will be reported in terms of groups of participants rather than as individual cases. In presentations and publications, participants' responses may be used in the form of quotations. However, no names or other identifying information will be included.

Those who will have access to your research records are the study personnel, the Institutional Review Board (IRB), and any other person, agency, or sponsor as required by law or contract or institutional responsibility. If these individuals were to access the data, your name would not be associated with it.

Finally, the CDC has asked researchers to share as much data from this study as we can with other researchers. We will share your data, without any information that could identify you, like your name or where you live, in a special database for other scientists who are doing research. We will only share de-identified data, in which research participants and schools will be identified by a number, and DMPS will be referred to as "a school district in a city in the Midwest" (or a similar variation). Sharing data helps scientists learn new and important things more quickly. Any scientists interested in using your data would have to put in a special request, promise to keep the data safe, and promise not to try to learn research participants' identities. We cannot remove your data if you change your mind because the data is anonymous. In summary, you are agreeing for your de-identified data (no names, etc.) to be put together with other people's data to be shared in a database by saying you want to be in this study. This sharing is not sharing your information for future research. It is only sharing anonymous/deidentified data from this specific study.

**Certificate of Confidentiality.** You should also know that we have a Certificate of Confidentiality from the Federal Government. This means that if someone came to us and asked for information about participants in this project, we could use this Certificate to refuse to give them information. This Certificate is to help us protect your privacy, but it does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you give your written consent to someone to receive research information, then we may not use the Certificate to withhold information.

**Public Information About this Study.** Clinical Trials.gov is a website that provides information about federally and privately supported clinical trials. A description of this clinical trial will be available (<a href="https://www.ClinicalTrials.gov">https://www.ClinicalTrials.gov</a>) as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.



What are the possible risks of being in this research study? The risks to participation are minimal. Sometimes when talking about topics like sex trafficking, people may feel sad, anxious, or awkward. However, you will be given a list of resources of places to go in the Des Moines area that may be helpful to you and/or the students you work with.

What are the possible benefits to you? You may not benefit from being in this project. However, some people tell us that they enjoy participating in research and like to share their ideas to help other people and their community.

What are the possible benefits to other people? The benefits to society include a better understanding of how to prevent sex trafficking of teens.

**What will being in this research study cost you?** There is no cost to you to be in this research study.

**Will you be compensated for being in this research study?** We will do a drawing for 5, \$100 incentives. We expect about 100 school personnel in the district to participate so each person has a 5% chance of winning an incentive. We will do the drawings within a few months of when you start this project. The person doing the drawing will be a researcher at UNL. They will do the drawing using a computer program to make sure it is fair and accurate. If you win an incentive, you will be asked to fill out a form saying you got the money. However, your survey answers will not be connected to the form confirming receipt of the incentive.

**How will information about you be protected?** If a physical copy of a research record is collected, it will be stored in a locked cabinet in the Project LIVE office until it is processed in a digital format. All paper copies will be destroyed following a muti-staff confirmation that records have been converted. The research records will be securely stored electronically through University-approved methods and will only be seen by the research team and/or those authorized to view, access, or use the records during and after the study is complete.

What are your rights as a research subject? You may ask any questions about this research and have those questions answered before agreeing to participate in or during the study. You can stop participating at any time and can choose not to answer any questions and still be eligible for compensation. You can decide if you want to be in the study or not. You can also stop participating ("withdraw") at any time before, during, or after the research begins for any reason. Deciding not to be in this research study, or deciding to withdraw, will not affect your relationship with the investigator, UNL, or DMPS.

Who should you contact if you have questions or concerns about this research project? If you have questions about this project, you can contact Dr. Katie Edwards, the principal investigator, by email (ProjectLIVE@unl.edu) or phone (515-410-6536). You can



also contact the Institutional Review Board (IRB) at UNL if you have questions about your rights as a participant or if you have concerns about this project at 402-472-6965 or irb@unl.edu.

**Documentation of informed consent.** You are voluntarily deciding whether or not to be in this research study. Signing this form means that (1) you have read and understood this consent form, (2) you have had the consent form explained to you, (3) you have had your questions answered, and (4) you have decided to be in the research study.

You can download a copy of this consent form to keep at <a href="https://cyfs.unl.edu/academies-bureaus/ivrl/current-projects/rts.php">https://cyfs.unl.edu/academies-bureaus/ivrl/current-projects/rts.php</a>

| Do you agree to participate? YES |
|----------------------------------|
| NO |
| Your Name: |
| School you work at: |
| Your Signature: |
| Date: |
| Your Email: |
| Your Phone Number: |

<sup>\*</sup>Contact information is collected ONLY to get you the gift card if you win the raffle. We will never share this.